CLINICAL TRIAL: NCT03491657
Title: Virtual Reality Analgesia for Pediatric Burn Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 71011-GAL
Record Dates: First submitted 2018-03-10; First posted 2018-04-09 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-03

CONDITIONS: Pain, Acute
Keywords: virtual reality pain; opioid; pediatric burn; wound care
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: Within-subject design with repeated measures, with random assignment to initial treatment.
Masking Description: Blinding can be challenging in behavioral studies. To help control for demand characteristics, the current study uses an active comparator "music distraction" vs. the experimental treatment condition "immersive virtual reality".
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality distraction (Yes VR) (Experimental): In addition to their standard pain medications, patients will play a virtual realty game named SnowWorld during some portions of their burn wound cleaning procedure, on each study day.
  Interventions: Behavioral: virtual reality distraction (Yes VR)
- music distraction (No VR condition) (Active Comparator): In addition to their standard pain medications, patients will listen to music during comparable portions of their burn wound cleaning procedure, on each study day.
  Interventions: Behavioral: music distraction (No VR)

INTERVENTIONS:
Behavioral: virtual reality distraction (Yes VR)
  Arms: virtual reality distraction (Yes VR)
Behavioral: music distraction (No VR)
  Arms: music distraction (No VR condition)

SUMMARY:
Many children with large severe burns report severe pain during burn wound cleaning. The current study explores whether adjunctive immersive Virtual Reality distraction may help reduce the intensity of pain experienced by children during burn wound cleaning by taking the patient's mind off their pain.

DETAILED DESCRIPTION:
All patients always receive their usual pain medications. Using a within-subjects, within-wound care design, in the current study, pediatric patients being treated for severe burn injuries will receive music distraction during some portions of their wound care (active comparator condition), and they will receive what we predict will be an unusually strong distraction, immersive virtual reality (the experimental treatment) during other comparable portions of the same wound cleaning sessions. During virtual reality, each patient will look into virtual reality goggles, and will play a simple cartoon-like virtual reality game SnowWorld during burn wound cleaning. After each wound care session, the patient will rate how much pain they experienced during wound care during No VR (music only) compared to how much pain they experienced during wound care during virtual reality, on each study day, for up to 10 study days per patient. Treatment order randomized.

ELIGIBILITY:
Inclusion criteria:

* Compliant and able to complete subjective evaluations,
* A minimum of 10% of total burned surface area,
* No history of psychiatric (DSM-III-R Axis I) disorder(s),
* Not demonstrating delirium, psychosis or any form of organic brain disorder,
* Able to communicate verbally in English or Spanish,
* Admitted to UTMB/Shriners, 6-17 years of age.

Exclusion criteria:

* No wound cleaning sessions required.
* Less than 10% of total burned surface area.
* History of psychiatric (DSM-III-R Axis I) disorder(s).
* Demonstrating delirium, psychosis or organic brain disorder.
* Unable to communicate verbally in English or Spanish.
* History of significant cardiac, endocrine, neurologic, metabolic, respiratory, gastrointestinal, or genitourinary impairment.
* Receiving prophylaxis for alcohol or drug withdrawal,
* Developmental disability, Younger than 6 years; older than 17 years,
* Burns of eyes, eyelids or face so severe they preclude the use of VR,
* Worst pain intensity of less than 5 on a 0 to 10 scale, during baseline No VR wound care Day 1.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2014-03-13 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
"Worst Pain" rating of pain intensity during Music vs. during VR | measured after burn wound care on each study day for up to 10 study days per patient
  worst pain during wound care. This single question measures the sensory component of pain during wound care. Patients will rate their "worst pain" during burn wound care. on a zero to ten scale, where zero is "no pain at all " and 10 is "excruciating pain". Lower scores represent better outcome. No subscales.

SECONDARY OUTCOMES:
Graphic Rating Scale "Time spent thinking about pain" during Music vs. during VR | measured after burn wound care on each study day for up to 10 study days per patient
  This single question measures the Cognitive component of pain during wound care. Patients will rate how much time they spent thinking about pain during burn wound care, on a zero to ten scale, where zero is "no time at all" and 10 is "the entire time". Lower scores represent better outcome. No subscales.
Graphic Ratings Scale measure of pain unpleasantness during Music vs. during VR | measured after woundcare on each study day for up to 10 study days per patient
  This single question measures the emotional component of pain. On a scale from zero to ten, where zero is "not unpleasant at all", 10 is "excruciatingly unpleasant". Lower scores represent better outcome. No subscales.
Graphic Rating Scale "Fun" during Music vs. during VR | measured after wound care on each study day for up to 10 study days per patient
  This single question measures positive affect during burn wound care. On a zero to ten scale, where zero is no fun at all and 10 is extremely fun. Higher scores represent better outcome. No subscales.
Graphic Rating Scale Satisfaction with pain management during Music vs. during VR | Measured after wound care on Study Day 1.
  This single question measures how satisfied the patient is with how well their pain was controlled during burn wound care. Higher scores represent better ourcomes. No subscales
Child Health Questionnaire | measured at 0, 9 months and 12 month followup visits
  Child Health Questionnaire The Child Health Questionnaire (CHQ) is a family of generic QOL instruments. The CHQ includes 87 scales that consider the effects of children's health on family functioning, and specific scales such as behavior and self-esteem. The CHQ measures 14 unique physical and psychosocial concepts. Questionnaires will be self-completed by the outpatients or parents, or both. Raw scores will converted to scaled scores from zero to 100. Higher scores indicate better health and better quality of life outcome.

OTHER OUTCOMES:
Sullivans Pain Catastrophizing Scale for Children (Crombez et al., 2003). | measured on Study day 1
  High catastrophizers are people who have unusually negative emotions and pessimistic beliefs about their ability to deal with the upcoming pain. Higher scores indicate worse outcome. 13 items, ratings from zero to 5 per item, 65 total points possible, 6 items measure helplessness, 3 items measure magnification, 4 items measure rumination subscores = 0-30 for helplessness, 0-15 for magnification, 0-20 for rumination. The PCS total score is calculated by summing the 13-item responses, and provides a good index of the catastrophizing construct through the inclusion of highly correlated subscales of helplessness, rumination, and magnification. Higher scores on the PCS are indicative of greater pain-related catastrophizing.

CONTACTS AND LOCATIONS:
Overall Officials: Walter J Meyer, MD, Principal Investigator — UTMB/Shriners
Locations (1):
- Shriners Hospital for Children; Shriners Burns Hospital, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared with other researchers. Any data shared with other researchers will be in unidentifiable form.

REFERENCES:
- [Background] Hoffman HG, Chambers GT, Meyer WJ 3rd, Arceneaux LL, Russell WJ, Seibel EJ, Richards TL, Sharar SR, Patterson DR. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann Behav Med. 2011 Apr;41(2):183-91. doi: 10.1007/s12160-010-9248-7. PMID 21264690
- [Background] Crombez G, Bijttebier P, Eccleston C, Mascagni T, Mertens G, Goubert L, Verstraeten K. The child version of the pain catastrophizing scale (PCS-C): a preliminary validation. Pain. 2003 Aug;104(3):639-646. doi: 10.1016/S0304-3959(03)00121-0. PMID 12927636
- See also: www.vrpain.com — http://www.vrpain.com